CLINICAL TRIAL: NCT05913557
Title: Targeting the Transdiagnostic Mechanism of Performance Monitoring and Overcontrol in Adolescence: Adaptation and Feasibility
Brief Title: Radical Openness for Adolescents Pilot
Acronym: ROA
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201912169
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Anorexia Nervosa; Obsessive-Compulsive Disorder; Social Phobia; Depression, Anxiety
MeSH Terms: conditions — Anorexia Nervosa; Obsessive-Compulsive Disorder; Phobia, Social; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants were either in a healthy group that did not receive treatment but did complete a baseline assessment or in one of two clinical groups. The first clinical group completed a baseline assessment, received 4 months of Radically Open Dialectical Behavior Therapy (RO DBT) treatment, then completed a follow-up assessment. The non-treatment clinical received no treatment (but could complete any other ongoing treatment as usual (TAU) treatment) and completed a baseline assessment and a subset also completed a follow-up assessment.
Masking Description: Participants self-selected to receive the therapy or not receive the therapy. Researchers and providers were also made aware of treatment group as they would then set up assessments and first treatment session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment Group (Experimental): Participants completed a baseline assessment, received 4 months of RO DBT therapy, then completed a follow-up assessment.
  Interventions: Behavioral: Radically Open Dialectical Behavior Therapy (RO DBT)
- No Treatment Group (No Intervention): Participants completed baseline assessment but did not receive treatment. A small subset also completed a follow-up assessment.
- Healthy Controls (No Intervention): Participants completed baseline assessment but did not receive treatment.

INTERVENTIONS:
Behavioral: Radically Open Dialectical Behavior Therapy (RO DBT) — Radically Open Dialectical Behavior therapy (RO DBT) is a type of cognitive behavioral therapy developed by Dr. Thomas Lynch for disorders of emotional overcontrol. RO DBT is a treatment indicated for patients across multiple psychiatric disorders, including diagnoses of chronic depression, treatment resistant anxiety disorders, anorexia nervosa, autism spectrum disorders, and avoidant, paranoid, and obsessive-compulsive personality disorders.
  Arms: Treatment Group

SUMMARY:
Heightened performance monitoring and overcontrol (HPM/OC) is characterized by inflexibility, a need for control, perfectionism, anxious apprehension and high error monitoring. HPM/OC is a cross-diagnostic (transdiagnostic) characteristic occurring across multiple forms of psychiatric illness that emerge in adolescence, including anorexia nervosa (AN), obsessive compulsive disorder (OCD) and social anxiety disorder. This study characterizes behavioral and neural HPM/OC in healthy adolescents and adolescents with disorders characterized by HPM/OC, including AN and related eating disorders and anxiety, depressive and obsessive compulsive disorders. We then examine feasibility of a novel treatment for HPM/OC in adolescents, examining recruitment feasibility, exploration of the mechanism of HPM/OC and examining whether treatment is able to target neural and behavioral HPM/OC.

DETAILED DESCRIPTION:
Eligible patient (n=30) and healthy (n=30) adolescents and young adults will attend a baseline session where they will undergo an ERP neural assessment and fill out questionnaires. 8 patient participants interested in participating in a 4 month free RO DBT therapy trial will participate in weekly individual and skills class sessions. At the end of this 4 months, they will complete a second follow-up session where they will undergo an event related potential (ERP) neural assessment and fill out questionnaires. 8 of the remaining 30 patient participants who do not want to complete the free therapy trial will have the option to return for a second follow-up session where they will undergo an ERP neural assessment and fill out questionnaires while undergoing treatment as usual (outside of therapy trial).

ELIGIBILITY:
Inclusion Criteria:

Adolescents with HPM/OC: Female adolescents and young adults with AN and related eating disordered pathology and other disorders of HPM/OC. Inclusion criteria include ages 13-21, female gender, and must be characterized by elevated dimensional HPM/OC. Inclusion criteria also require a psychiatric disorder and/or impairment related to HPM/OC, including a diagnosis of AN, related eating disordered pathology related to AN that is characterized by HPM/OC (Eating disorder not otherwise specified; EDNOS; with high HPM/OC),and/or a diagnosis of a related disorder characterized by HPM/OC, namely obsessive compulsive disorder (OCD) or social anxiety disorder. Importantly, not only psychiatric illness, but psychiatric illness characterized by HPM/OC is required. Participants will not be excluded due to medication status. Other inclusion include: for adolescents younger than 17, the consent and participation of a legal caregiver. Other inclusion include if participating in therapy beyond baseline session: living in the St. Louis region (to attend sessions) and willingness to have RO DBT-A as only psychosocial treatment engaged in (medication treatment may continue).

Healthy adolescents: Female adolescents and young adults age 13-21 matched to patient sample on age and gender (all females). Inclusion criteria: no diagnosis of disorders of HPM/OC, including AN and related eating disordered pathology, OCD, or social anxiety disorder, ability to complete the EEG and baseline session, and scores below the clinical cut-off on a questionnaire, the Youth Self Report (YSR).

Exclusion Criteria:

Adolescents with HPM/OC: Exclusion criteria include: male gender, outside age range, significant developmental or cognitive delays, seizure or other major neurological disorder, severe head injury, inability to understand, speak and read English sufficiently (both adolescent and caregiver if under age 18).

Healthy adolescents: Exclusion criteria: male gender, outside age range, significant developmental or cognitive delays, seizure or other major neurological disorder, severe head injury, inability to understand, speak and read English sufficiently (both adolescent and caregiver if under age 18), or disorder of AN, OCD, Social Anxiety Disorder.

Ages: 13 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Changes in error-related negativity (ERN) amplitudes | Baseline (all groups), 4 months (treatment group, no treatment group [subset completing follow-up])
  ERN data is obtained during electroencephalogram (EEG) sessions during which participants engage in several behavioral tasks. These tasks include Flankers (participant must quickly press an arrow key that corresponds to the center arrowhead depicted on the screen)
Changes in scores on Overcontrol Youth Checklist (OCYC) | Baseline (all groups), 4 months (treatment group, no treatment group [subset completing follow-up])
  The OCYC is a validated self-report checklist that assesses levels of hyper-performance monitoring and overcontrol. The youth is asked to respond yes/no to a variety of personality-based questions. A total score is generated, as well as a frustration/rigidity score and a social concern/perfectionism score.
Changes in scores on Adolescent Over- and Under-control Trait Measure (OUT'M) | Baseline (all groups), 4 months (treatment group, no treatment group [subset completing follow-up])
  The OUT'M is a validated self-report checklist that assesses levels of overcontrol as well as undercontrol. Youths are asked to rate themselves on a variety of personality traits using a scale from 0-6. Overcontrol and undercontrol scores are generated.
Changes in Behavioral Reward Responding using the Temporal Experience of Pleasure Scale (TEPS), including the anticipatory and consummatory subscales | Baseline (all groups), 4 months (treatment group, no treatment group [subset completing follow-up])
  The TEPS is an 18-item measure, rated from one ("very false for me") to six ("very true for me"; α = 0.89). Examples of items include "I look forward to a lot of things in my life" (anticipatory) and "I enjoy taking a deep breath of fresh air when I walk outside" (consummatory).
Changes in Reward Positivity (RewP) amplitudes | Baseline (all groups), 4 months (treatment group, no treatment group [subset completing follow-up])
  RewP data is obtained during electroencephalogram (EEG) sessions during which participants engage in a behavioral task of opening a door and receiving a small amount of money to win if they open the correct door, or lose a small amount of money if they do not open the 'correct' door. The RewP is measured by examining neural response to winning money subtracting out the neural response to losing money.

SECONDARY OUTCOMES:
Changes in disruptive eating symptomology using Eating Disorder Examination-Questionnaire (EDE-Q) | Baseline (all groups), 4 months (treatment group, no treatment group [subset completing follow-up])
  The EDE-Q is a self-report measure of eating disorder pathology for the last 28 days. It is a 36-item, 7-point scale (Fairburn & Beglin, 1994). The resulting global score (α = 0.83), and four subscales, are comprised of item averages which, when over 4, indicate clinically significant eating pathology.
Changes in anxious symptomology using Screen for Child Anxiety Related Disorders (SCARED) | Baseline (all groups), 4 months (treatment group, no treatment group [subset completing follow-up])
  The SCARED is a 41-item scale (α = 0.90) rated from zero ("Not True or Hardly Ever True") to two ("Very True or Often True"). Summed total scores (α = 0.90) over 25 indicate clinically significant anxiety.
Changes in functional impairment using Pediatric Quality of Life Enjoyment and Satisfaction Questionnaire (PQLES-Q) | Baseline (all groups), 4 months (treatment group, no treatment group [subset completing follow-up])
  The PQLES-Q is a 15-item scale, with items rated from one ("Very Poor") to six ("Very Good") where the first 14 items are summed for a total score and the last item is a self-reported global measure (α = 0.93). Higher scores indicate higher satisfaction and enjoyment.
Changes in social impairment using Social Connectedness Scale (SCS) | Baseline (all groups), 4 months (treatment group, no treatment group [subset completing follow-up])
  The SCS is an 8-item measure, rated from one ("Agree") to six ("Disagree") and summed, with higher scores indicating more social connectedness (α = 0.91). An example item from the SCS is "I feel so distant from people".
Changes in depressive symptomology using Child Depression Inventory (CDI) | Baseline (all groups), 4 months (treatment group, no treatment group [subset completing follow-up])
  The CDI is a 27-item scale rated from 0 to 2 and summed to create a total score. The suicidality question was omitted, yielding 26 questions. The T-score of the total score was used (α = 0.92).

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

DOCUMENTS (1):
  • Informed Consent Form (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT05913557/ICF_000.pdf